CLINICAL TRIAL: NCT06551519
Title: A Non-interventional Study Evaluating Clinical Utility and Implications on Improved Patient Management of Serum Neurofilament as a Prognostic Marker for Disease Activity in Patients With Relapsing Multiple Sclerosis (FILAXOS)
Brief Title: A Non-interventional Study Evaluating Clinical Utility and Implications on Improved Patient Management of Serum Neurofilament as a Prognostic Marker for Disease Activity in Patients With Relapsing Multiple Sclerosis
Acronym: FILAXOS
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GDE04
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; MS; Ofatumumab; NIS; Germany
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Ofatumumab: Patients who have received treatment with category 1 DMTs and decided to switch to ofatumumab
  Interventions: Other: ofatumumab
- Category 1 DMTs: Patients who continued with DMT category 1 treatment. According to local treatment guidelines, DMT category 1 include dimethylfumarate/diroximelfumarate, glatirameroids, Interferon beta and teriflunomide.
  Interventions: Other: DMT category 1

INTERVENTIONS:
Other: ofatumumab — This is an observational study. There is no treatment allocation. The decision to initiate ofatumumab will be based solely on clinical judgement.
  Groups: Ofatumumab
Other: DMT category 1 — This is an observational study. There is no treatment allocation. The decision to continue their current DMT will be based solely on clinical judgement.
  Groups: Category 1 DMTs

SUMMARY:
This is a prospective, multicenter, observational, non-interventional study (NIS) in patients with Multiple Sclerosis (MS) and routinely assessed serum neurofilament light (sNfL) values in Germany

DETAILED DESCRIPTION:
Prospective, primary data will be collected from patients with sNfL outcomes in the context of switching to ofatumumab or continuing their current therapy. Data collection will cover a maximum period of 24 months.

The observational period will not be dictated by the protocol. Baseline and follow-up visits will take place at a frequency defined as per Investigator´s discretion following clinical routine. The diagnostic or monitoring procedures are only those ordinarily applied to therapeutic strategy and routine clinical care. During the observation phase of the study, data will be collected according to standard of care as recommended by KKNMS (Competence Network Multiple Sclerosis in Germany).

Eligible participants for the study are patients who have received treatment with category 1 DMTs and those who have included sNfL into their treatment decision-making process. These patients have the option to either continue their current DMT or switch to ofatumumab. According to local treatment guidelines, DMT category 1 include dimethylfumarate/diroximelfumarate, glatirameroids, Interferon beta and teriflunomide. The decision to switch to ofatumumab or to continue the current DMT category 1 therapy must be made by the treating physician independently of the decision to enroll the patient in the study.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all the following criteria:

1. Written informed consent must be obtained before participation in the study.
2. RMS patients aged 18 or older.
3. Treated in label with EU-approved DMTs for MS category 1 according to current guidelines (Hemmer et al 2023) for at least the last 3 months.
4. Presence of a sNfL test result from a commercially available test not older than 3 months.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study:

1. Patients being treated outside of the approved label of the respective DMT.
2. Simultaneous participation in any interventional study or simultaneous participation in another Novartis-sponsored non-interventional study with ofatumumab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients currently treated with a DMT category 1 prior to study start and receive sNfL measurements
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-11-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with high serum neurofilament light (sNfL) levels | Up to 24 months
  Proportion of patients with high serum neurofilament light (sNfL) levels within 24 months of observation

SECONDARY OUTCOMES:
sNfL use as a biomarker for Multiple Sclerosis disease activity in clinical practice | Up to 24 months
  Description of perception, utility, frequency of serum neurofilament light (sNfL) measurements and clinical consequences initiated by the treating physician in clinical routine care setting
Proportion of patients demonstrating radiological and / or clinical activity | Up to 24 months
  Proportion of patients demonstrating radiological (number of new/enlarging T2 lesions, number of Gadolinium-positive T1 lesions) and / or clinical activity (MS relapse, confirmed disability progression) at Baseline and throughout the study also in context with sNfL level.
Proportion of patients with no evidence of disease activity (NEDA) | Baseline, month 12 and month 24
  Proportion of patients with NEDA at 12 and 24 months as compared to Baseline also in context with sNfL level.
Proportion of patients demonstrating NEDA 3 and its individual components at 24 months as compared to Baseline | Baseline, 24 months
  NEDA is defined by no confirmed multiple sclerosis relapse, no new or enlarging T2 lesions, no Gadolinium-positive T1 lesions, and no six-month confirmed disability worsening.
Proportion of patients perceived as clinically stable depending on sNfL level | Up to 24 months
  Proportion of patients perceived as clinically stable depending on sNfL level
Multiple sclerosis impact scale 29 (MSIS-29) | Up to 24 months
  The Multiple Sclerosis Impact Scale version 2 will be used to assess health-related quality of life. MSIS-29 is a 29-item, self-administered questionnaire that includes two domains, physical and psychological. Responses are captured on a 4-point scale ranging from "not at all" (1) to "extremely" (4), where higher scores reflect greater impact on day-to-day life.
Fatigue questionnaire: Fatigue Scale for Motor and Cognitive Functions (FSMC) | Up to 24 months
  FSMC consists of 20 items (10 for cognitive fatigue [FSMCcog] and 10 for motor fatigue [FSMCmot]) with 1-5 points per item. The total possible score ranges from 20-100 points. A sum score of ≥43 is categorized as mild fatigue, ≥53 as moderate fatigue and ≥63 as severe fatigue.
EuroQol- 5 Dimension (EQ-5D) score | Up to 24 months
  This patient questionnaire is a generic multidimensional measure of health-related quality of life (EuroQol 1990). The five domains of mobility, ability to take care of oneself, everyday activities, pain/discomfort and anxiety/depression are considered. For each dimension, the most appropriate answer is selected from three given possibilities (1=no problem, 2=moderate problem, 3=big problem). In addition, the patient marks the current state of health on a scale from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
Number of participants using Ekiva MS App | Up to 24 months
  Change in satisfaction scores and evaluation of improvement of patient-physician dialogue and Multiple Sclerosis patient management
Treatment Satisfaction Questionnaire for Medication (TSQM) score | Up to 24 months
  The TSQM Version 1.4 comprises 14 items across four domains focusing on effectiveness (3 items), side effects (5 items), convenience (3 items), and global satisfaction (3 items) of the medication over the previous 2-3 weeks, or since the subject´s last use. With the exception of item 4 (presence of side effects; yes or no), all items have 5 or 7 responses, scored from 1 (least satisfied) to 5 or 7 (most satisfied). The 7-item scales had a non-neutral midpoint, such that there were more positive response options than negative response options, to allow precise information to be obtained at the upper end of the score distribution. Item scores are summarized to give four domain scores, which are in turn transformed to a scale of 0-100.
Reasons for and proportion of patients switching from current DMTs to ofatumumab | Up to 24 months
  Reasons for and proportion of patients switching from current DMTs to ofatumumab depending on sNfL level
Proportion of missed ofatumumab doses within one year, | Month 12
  Proportion of missed ofatumumab doses within one year, defined as the difference between number of planned doses and number of administered doses.
Proportion of patients who continue to receive their initial treatment | Month 12 and month 24
  Proportion of patients who continue to receive their initial treatment (ofatumumab or DMT category 1)
Reasons for, number of and duration of treatment interruptions and discontinuations. | Up to 24 months
  Reasons for and number of treatment interruptions and discontinuations.
Duration of treatment interruptions and discontinuations. | Up to 24 months
  Duration of treatment interruptions and discontinuations.
Characterization of patient subgroups with and without 100% adherence | Month 12
  Patients with matching number of planned doses and number of administered doses within 1 year (eg, previous experience with sub-cutaneous therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (89):
- Germany (89):
  - Novartis Investigative Site, Albstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Hettingen, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Schwetzingen, Baden-Wurttemberg
  - Novartis Investigative Site, Bamberg, Bavaria
  - Novartis Investigative Site, Neuburg an der Donau, Bavaria
  - Novartis Investigative Site, Untermeiting, Bavaria
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Bad Homburg, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Meerbusch, North Rhine-Westphalia
  - Novartis Investigative Site, Siegen, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Görlitz, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Altenburg, Thuringia
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Mühlhausen, Thuringia
  - Novartis Investigative Site, Aalen
  - Novartis Investigative Site, Altenholz
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Backnang
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bergneustadt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bogen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dillingen Saar
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisleben Lutherstadt
  - Novartis Investigative Site, Eltville
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Herford
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Höxter
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Katzenelnbogen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Merzig
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Salzatal
  - Novartis Investigative Site, Schiltach
  - Novartis Investigative Site, Schwalmstadt-Treysa
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Sundern Hachen
  - Novartis Investigative Site, Tirschenreuth
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Weil der Stadt
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wolfenbüttel
  - Novartis Investigative Site, Wolfratshausen

IPD SHARING:
Plan to Share IPD: No